CLINICAL TRIAL: NCT05718336
Title: Atrial Fibrillation Trial To Eliminate Risk-factors
Acronym: AFTTER
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202003090RINA
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Integrated care — multi-discipline care program

SUMMARY:
The goal of this prospective-enrolling cohort study is to test and observe the effect of an integrated multi-discipline care program in patients with atrial fibrillation. The main questions it aims to answer are:

1. to understand the baseline characteristics and to explore the occult risk factors of the patients with AF;
2. to monitor the treatment efficacy of the patients undergoing integrated care and potentially concur the clinical obstacles that prevent the best care for patients with AF.

Participants will be treated by an integrated multi-discipline team that led by an electro-physiologist.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a heart condition that potentially leads to heart failure and ischemic stroke. The prevalence of AF is increasing due to aging population and improved treatment in other cardiovascular field. This study is to execute integrated multi-discipline care in a tertiary hospital, and to observe the effect and the obstacle that the program might ensue.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old, who have been diagnosed with atrial fibrillation by a cardiologist with an electrocardiogram

Exclusion Criteria:

1. Unable to complete the initial assessment and cooperate with the tracker
2. Those who refuse to sign the subject's consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with documented atrial fibrillation, either paroxysmal, persistent, or permanent.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
AF burden | 0~24 months
  The duration in AF on 14-day ECG monitor (percent)

SECONDARY OUTCOMES:
MACE, major adverse cardiovascular event | 0~24 months
  ischemic heart disease with acute coronary syndrome, stroke (either ischemic or hemorrhagic stroke), cardiovascular death, and all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chieh Yu, MD.PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospita, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No